CLINICAL TRIAL: NCT02966665
Title: Vascular Function in Health & Disease: Rehabilitation for Hypertension; Exercise and Skeletal Muscle Afferent Feedback
Brief Title: : Vascular Function in Health and Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Russell Richardson (Other)
Responsible Party: Sponsor-Investigator, Russell Richardson, Ph.D., University of Utah
Organization: University of Utah (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB_00030810
Record Dates: First submitted 2016-10-19; First posted 2016-11-17 (Estimated); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease; Pulmonary Artery Hypertension; Heart Failure; Hypertension
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Familial Primary Pulmonary Hypertension; Heart Failure; Hypertension | interventions — omega-N-Methylarginine; Ascorbic Acid; Vitamin E; Thioctic Acid; cyclo(Trp-Asp-Pro-Val-Leu); fexofenadine; Ranitidine; Angiotensin I; Valsartan; Acetylcholine; Nitroprusside; Norepinephrine; Phentolamine; mitoquinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Healthy Young Volunteers (18-30 years) (Experimental): Healthy volunteers between the ages of 18 and 30 years with no diseases or conditions that would affect their participation in the study, administered various treatments to assess their effect on blood flow and metabolic demand of tissues under wide-ranging conditions, including Maximum Exercise Tests, L-NMMA, Vitamin C, Vitamin E, α-Lipoic Acid, L-Ascorbate, BQ-123, Fexofenadine, Ranitidine, Angiotensin-II, Valsartan, Acetylcholine, Sodium Nitroprusside, Norepinephrine, Phentolamine and MitoQ.
  Interventions: Other: Maximum Exercise Tests; Drug: BH4, L-NMMA, Vitamin C, Vitamin E, α-Lipoic Acid and L-Ascorbate; Drug: BQ-123; Drug: Fexofenadine, Ranitidine; Other: Angiotensin-II, Valsartan; Drug: Acetylcholine, Sodium Nitroprusside, Angiotensin-II, Norepinephrine, Phentolamine; Drug: BQ-123, MitoQ, BH4
- Healthy Older Controls (over 65 years) (Experimental): Healthy volunteers 65 years of age or older with no diseases or conditions that would affect their participation in the study, administered various treatments to assess their effect on blood flow and metabolic demand of tissues under wide-ranging conditions, including Maximum Exercise Tests, L-NMMA, Vitamin C, Vitamin E, α-Lipoic Acid, L-Ascorbate, BQ-123, Fexofenadine, Ranitidine, Angiotensin-II, Valsartan, Acetylcholine, Sodium Nitroprusside, Norepinephrine, Phentolamine and MitoQ.
  Interventions: Other: Maximum Exercise Tests; Drug: BH4, L-NMMA, Vitamin C, Vitamin E, α-Lipoic Acid and L-Ascorbate; Drug: BQ-123; Drug: Fexofenadine, Ranitidine; Other: Angiotensin-II, Valsartan; Drug: Acetylcholine, Sodium Nitroprusside, Angiotensin-II, Norepinephrine, Phentolamine; Drug: BQ-123, MitoQ, BH4
- Coronary Angiography patients (Experimental): Patients undergoing routine coronary angiography, but who do not require intracoronary procedures or have history of myocardial disease, administered various treatments to assess their effect on blood flow and metabolic demand of tissues under wide-ranging conditions, including Maximum Exercise Tests, L-NMMA, Vitamin C, Vitamin E, α-Lipoic Acid, L-Ascorbate, BQ-123, Fexofenadine, Ranitidine, Angiotensin-II, Valsartan, Acetylcholine, Sodium Nitroprusside, Norepinephrine, Phentolamine and MitoQ.
  Interventions: Other: Maximum Exercise Tests; Drug: BH4, L-NMMA, Vitamin C, Vitamin E, α-Lipoic Acid and L-Ascorbate; Drug: BQ-123; Drug: Fexofenadine, Ranitidine; Other: Angiotensin-II, Valsartan; Drug: Acetylcholine, Sodium Nitroprusside, Angiotensin-II, Norepinephrine, Phentolamine; Drug: BQ-123, MitoQ, BH4
- Chronic Obstructive Pulmonary Disease patients (Experimental): Patients diagnosed with mild to moderate COPD, but not severe COPD patients, administered various treatments to assess their effect on blood flow and metabolic demand of tissues under wide-ranging conditions, including Maximum Exercise Tests, L-NMMA, Vitamin C, Vitamin E, α-Lipoic Acid, L-Ascorbate, BQ-123, Fexofenadine, Ranitidine, Angiotensin-II, Valsartan, Acetylcholine, Sodium Nitroprusside, Norepinephrine, Phentolamine and MitoQ.
  Interventions: Other: Maximum Exercise Tests; Drug: BH4, L-NMMA, Vitamin C, Vitamin E, α-Lipoic Acid and L-Ascorbate; Drug: BQ-123; Drug: Fexofenadine, Ranitidine; Other: Angiotensin-II, Valsartan; Drug: Acetylcholine, Sodium Nitroprusside, Angiotensin-II, Norepinephrine, Phentolamine; Drug: BQ-123, MitoQ, BH4
- Pulmonary Arterial Hypertension patients (Experimental): Patients with idiopathic or heritable Group 1 pulmonary arterial hypertension, administered various treatments to assess their effect on blood flow and metabolic demand of tissues under wide-ranging conditions, including Maximum Exercise Tests, L-NMMA, Vitamin C, Vitamin E, α-Lipoic Acid, L-Ascorbate, BQ-123, Fexofenadine, Ranitidine, Angiotensin-II, Valsartan, Acetylcholine, Sodium Nitroprusside, Norepinephrine, Phentolamine and MitoQ.
  Interventions: Other: Maximum Exercise Tests; Drug: BH4, L-NMMA, Vitamin C, Vitamin E, α-Lipoic Acid and L-Ascorbate; Drug: BQ-123; Drug: Fexofenadine, Ranitidine; Other: Angiotensin-II, Valsartan; Drug: Acetylcholine, Sodium Nitroprusside, Angiotensin-II, Norepinephrine, Phentolamine; Drug: BQ-123, MitoQ, BH4
- Heart Failure patients (Experimental): Patients with Class I - III New York Heart Association symptoms of Heart Failure who are not anemic or taking medications that affect blood clotting, administered various treatments to assess their effect on blood flow and metabolic demand of tissues under wide-ranging conditions, including Maximum Exercise Tests, L-NMMA, Vitamin C, Vitamin E, α-Lipoic Acid, L-Ascorbate, BQ-123, Fexofenadine, Ranitidine, Angiotensin-II, Valsartan, Acetylcholine, Sodium Nitroprusside, Norepinephrine, Phentolamine and MitoQ.
  Interventions: Other: Maximum Exercise Tests; Drug: BH4, L-NMMA, Vitamin C, Vitamin E, α-Lipoic Acid and L-Ascorbate; Drug: BQ-123; Drug: Fexofenadine, Ranitidine; Other: Angiotensin-II, Valsartan; Drug: Acetylcholine, Sodium Nitroprusside, Angiotensin-II, Norepinephrine, Phentolamine; Drug: BQ-123, MitoQ, BH4
- Hypertension patients (Experimental): Patients with chronic high blood pressure, but with less than severe hypertension, administered various treatments to assess their effect on blood flow and metabolic demand of tissues under wide-ranging conditions, including Maximum Exercise Tests, L-NMMA, Vitamin C, Vitamin E, α-Lipoic Acid, L-Ascorbate, BQ-123, Fexofenadine, Ranitidine, Angiotensin-II, Valsartan, Acetylcholine, Sodium Nitroprusside, Norepinephrine, Phentolamine and MitoQ.
  Interventions: Other: Maximum Exercise Tests; Drug: BH4, L-NMMA, Vitamin C, Vitamin E, α-Lipoic Acid and L-Ascorbate; Drug: BQ-123; Drug: Fexofenadine, Ranitidine; Other: Angiotensin-II, Valsartan; Drug: Acetylcholine, Sodium Nitroprusside, Angiotensin-II, Norepinephrine, Phentolamine; Drug: BQ-123, MitoQ, BH4

INTERVENTIONS:
Other: Maximum Exercise Tests — Graded exercise test to volitional exhaustion (stationary bike or treadmill), maximal handgrip test, maximal leg extension test, and maximal plantar flexion test.
Drug: BH4, L-NMMA, Vitamin C, Vitamin E, α-Lipoic Acid and L-Ascorbate — Catheter placement in femoral artery and femoral vein; resting measurements of blood pressure, heart rate and blood flow; flow mediated vasodilation test, passive leg movement test, exercise bouts, electromyography and exercise training regimen at baseline and following treatment with Nitric Oxide blockade via infusion of N-monomethyl-L-arginine (L-NMMA) (0.4 mg/kg/min), antioxidant cocktail (Vitamin C, Vitamin E, alpha-lipoic acid) ingestion, L-ascorbate injection, BH4 ingestion.
Drug: BQ-123 — Catheter placement in femoral artery and femoral vein; resting measurements of blood pressure, heart rate and blood flow; flow mediated vasodilation test and exercise bouts at baseline and following treatment with endothelin-1 receptor antagonist BQ-123 (D-tryptamine-D-aspartic acid-L-proline-D-valine-L-leucine).
Drug: Fexofenadine, Ranitidine — Catheter placement in femoral artery and femoral vein; resting measurements of blood pressure, heart rate and blood flow; flow mediated vasodilation test and exercise bouts at baseline and following treatment with Histamine H1 receptor antagonist fexofenadine (Allegra) and Histamine H2 receptor antagonist ranitidine (Zantac).
  Other Names: Allegra; Zantac
Other: Angiotensin-II, Valsartan — Catheter placement in femoral artery and femoral vein; resting measurements of blood pressure, heart rate and blood flow; flow mediated vasodilation test, muscle sympathetic nerve activity measurement, and exercise bouts at baseline and following treatment with Angiotensin-II receptor agonist (angiotensin-II) and antagonist Valsartan (Diovan).
  Other Names: Diovan
Drug: Acetylcholine, Sodium Nitroprusside, Angiotensin-II, Norepinephrine, Phentolamine — Catheter placement in femoral artery and femoral vein; resting measurements of blood pressure, heart rate and blood flow; flow mediated vasodilation test, muscle sympathetic nerve activity measurement; vasodilation with nitroglycerin followed by Angiotensin-II and Alpha Adrenergic blockade with infusions of Acetylcholine, Sodium Nitroprusside, Angiotensin-II, Norepinephrine and Phentolamine (Regitine).
  Other Names: Regitine
Drug: BQ-123, MitoQ, BH4 — Catheter placement in femoral artery and femoral vein and muscle biopsy; Nuclear Magnetic Resonance (NMR) scanning and exercise bouts at baseline and following treatment with BQ-123 with or without oral mitochondria-targeted antioxidant (MitoQ) or oral BH4.

SUMMARY:
Many control mechanisms exist which successfully match the supply of blood with the metabolic demand of various tissues under wide-ranging conditions. One primary regulator of vasomotion and thus perfusion to the muscle tissue is the host of chemical factors originating from the vascular endothelium and the muscle tissue, which collectively sets the level of vascular tone. With advancing age and in many disease states, deleterious adaptations in the production and sensitivity of these vasodilator and vasoconstrictor substances may be observed, leading to a reduction in skeletal muscle blood flow and compromised perfusion to the muscle tissue. Adequate perfusion is particularly important during exercise to meet the increased metabolic demand of the exercising tissue, and thus any condition that reduces tissue perfusion may limit the capacity for physical activity. As it is now well established that regular physical activity is a key component in maintaining cardiovascular health with advancing age, there is a clear need for further studies in populations where vascular dysfunction is compromised, with the goal of identifying the mechanisms responsible for the dysfunction and exploring whether these maladaptations may be remediable. Thus, to better understand the etiology of these vascular adaptations in health and disease, the current proposal is designed to study changes in vascular function with advancing age, and also examine peripheral vascular changes in patients suffering from chronic obstructive pulmonary disease (COPD), Sepsis, Pulmonary Hypertension, and cardiovascular disease. While there are clearly a host of vasoactive substances which collectively act to govern vasoconstriction both at rest and during exercise, four specific pathways that may be implicated have been identified in these populations: Angiotensin-II (ANG-II), Endothelin-1 (ET-1), Nitric Oxide (NO), and oxidative stress.

DETAILED DESCRIPTION:
Angiotensin-II (ANG-II) is the end-product of the renin-angiotensin cascade, and acts as a potent endogenous vasoconstrictor through binding to the angiotensin receptor (AT1) on arteriolar vascular smooth muscle. With advancing age, there is a notable decline in plasma renin activity accompanied by decrements in circulating ANG-II and an increase in AT1 receptor density. However, the functional consequence of this age-related adaptation of the renin-angiotensin system (RAS) on the peripheral circulation is not well understood. Likewise, in recent years it has become apparent that cardiovascular disease is a major cause of morbidity in COPD, which may be related to vascular dysfunction and associated adoption of a sedentary lifestyle. In these patients, changes in RAS activity have been linked to peripheral vascular dysfunction, with compelling evidence for improvements in peripheral oxygen use following angiotensin-converting enzyme (ACE) inhibition. Like the aging population, systematic studies evaluating AT1 receptor sensitivity and the efficacy of AT1 receptor blockade on peripheral hemodynamics have not been undertaken.

The ubiquitous substance nitric oxide (NO) is now recognized as a key pathway for endothelium-dependent vasodilation, with the bioavailability of NO serving as an indicator for overall vascular health. Cardiac risk factors have been shown to cause impairment in endothelial vasodilator function in both the peripheral and coronary arteries. Coronary vascular dysfunction is an important phase in atherogenesis and is associated with myocardial ischemia. Furthermore, peripheral vascular function has been linked to coronary vascular dysfunction which could have important clinical implications in terms of health screening. Impaired endothelium-dependent vasodilation has been associated with the elderly, patients with COPD, and most cardiovascular diseases including pulmonary hypertension, and heart failure (HF), though the functional consequence of this adaptation on peripheral blood flow regulation remains unclear. Thus, we propose the use of a compound which inhibits the enzyme responsible for NO production in endothelial cells, N-monomethyl-L-arginine (L-NMMA), to temporarily block production of NO and thus determine the importance of this pathway at rest and during physical activity. Additionally, we propose the use of acetylcholine (Ach) to determine endothelial-dependent vasodilation and sodium nitroprusside (SNP) and nitroglycerin (NTG) to determine the endothelial-independent vasodilation in the coronary arteries and the periphery. Oxidative stress associated with aging has been shown to reduce vascular function and antioxidant supplementation restores vascular function to levels that are indistinguishable from healthy young adults. The manner by which this improvement in vascular function occurs is not known by may be acting through a NO dependent mechanism.

Histamine has been reported to mediate sustained post-exercise vasodilation through histamine-1 (H1) and histamine-2 (H2) receptor activity, which results in a ~50% elevation in femoral artery blood flow (above resting levels) that lasts for more than 100 minutes after a single bout of moderate-intensity dynamic exercise. Vasodilation can be markedly reduced by giving either fexofenadine (Allegra, a selective H1-receptor antagonist) or ranitidine (Zantac, a selective H2-receptor antagonist). The combination of H1/H2 blockade abolishes ~80% of the post-exercise vasodilation seen after whole-body exercise such as cycling and this observation has been observed in multiple studies in young sedentary, recreationally active, and endurance trained men and women. The impact of histamine on the post-exercise vasodilatory response is substantial; however, the role of H1/H2 receptors in regulating skeletal muscle blood flow during exercise is unknown. Thus, we intend to investigate the role of H1/H2 receptors in the regulation of skeletal muscle blood during exercise as this may be an important pathway in age and disease related reductions in blood flow during exercise.

Exercise training and rehabilitation can be used as an alternative approach to combat the deleterious effects oxidative stress on aging and disease. An effective exercise training intervention can decrease sympathetic nervous system activity, improve arterial compliance and vascular endothelial function, and alter the pro- and antioxidant balance resulting in improved endogenous antioxidant defense mechanisms. Moreover, exercise training concomitantly improves musculoskeletal strength and function, glucose regulation and insulin sensitivity, cardiovascular function, body composition, blood chemistry (decreased triglyceride and cholesterol levels), and overall well-being. The physiologic effect of an exercise rehabilitation program in diseases such as COPD, and pulmonary arterial hypertension (PAH) is incompletely understood. However, recent studies suggest that exercise training in this patient population is well tolerated and associated with clinically significant physiologic improvements as well as improvements in various quality of life scores.

A unique feature of the proposed studies identified herein is the inclusion of a novel methodological approach to comprehensively evaluate the functional outcome of the proposed pharmacologic interventions. The recent development of a unique combination of nuclear magnetic resonance (NMR) techniques by members of our group enables near-simultaneous measurements of both muscle perfusion and metabolism in vivo. The arterial spin labeling (ASL) technique allows the measurement of both spatially and temporally resolved quantification of perfusion, while the kinetics of phosphocreatine (PCr) depletion and recovery provide high resolution measurements of muscle energetics. The interweaving of these imaging and spectroscopic modules provides the opportunity for determination of skeletal muscle perfusion and metabolism kinetics during and following the stress of physical exercise. Thus, this NMR-based approach, combined with direct measures of muscle fatigue, offers the potential to further define the individual and collective contribution of these variables to the attenuated limb blood flow in the elderly and in patients with COPD and PAH.

We propose that each of these pathways outlined above represent an avenue by which vascular function is compromised in the elderly and in patients with COPD, PAH and cardiovascular disease. However, because these pathways are not mutually exclusive, the proposed studies are designed to systematically evaluate hemodynamic responses to intra-arterial or intravenous administration of pharmacologic agents specific for the AT1 receptor (ANG-II and Diovan, AT1 agonist and antagonist, respectively), the Endothelin receptor Type-A (ETA receptor) (BQ-123, ETA antagonist), and the NO pathway (L-NMMA, Ach, and SNP) both before and after exercise training.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Young Volunteers: 18-30 years of age with no diseases or conditions that would affect their participation in the study
* Healthy Older Controls: volunteers 65 years of age or older with no diseases or conditions that would affect their participation in the study
* Coronary Angiography subjects: patients undergoing routine coronary angiography
* Chronic Obstructive Pulmonary Disease subjects: patients diagnosed with mild to moderate COPD
* Pulmonary Arterial Hypertension subjects: patients with idiopathic or heritable Group 1 pulmonary arterial hypertension
* Heart Failure subjects: patients with Class I, II or III New York Heart Association symptoms of Heart Failure
* Hypertension subjects: patients diagnosed with chronic high blood pressure

Exclusion Criteria:

* Severe COPD (use of supplemental oxygen, or have a one-second forced expiratory volume of less than 30% predicted)
* History of myocardial infarction
* History of percutaneous coronary revascularization
* History of coronary artery bypass grafting
* Unstable angina pectoris
* History of variant angina
* Ejection fraction < 50%
* Significant renal disease (Glomerular Filtration Rate < 50 mL/min/1.73m2)
* Subjects whose medical care or safety may be at risk from undergoing a Magnetic Resonance Imaging examination (e.g. pacemaker, metal implants, certain types of heart valves)
* Subject is pregnant
* Subject has physical ailments (other than COPD, PAH, HF, or hypertension) that would prevent them from study participation in the judgment of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2008-09; Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in Limb Blood Flow | Baseline and 1 hour
  Change in local limb blood flow as measured by ultrasound Doppler in units of milliliters per minute (mL/min) from baseline to up to 1 hour following study interventions

SECONDARY OUTCOMES:
Change in Blood Pressure | Baseline and 1 hour
  Change in local limb blood pressure measured in millimeters of mercury (mmHg) from baseline to up to 1 hour following study interventions
Change in Maximum Exercise Capacity | Baseline and 1 hour
  Change in maximal exercise capacity - handgrip strength measured by dynamometer in units of kilograms from baseline to up to 1 hour following study interventions
Change in Peak Rate of Mitochondrial Adenosine Triphosphate (ATP) Synthesis | Baseline and 1 hour
  Change in muscle peak rate of mitochondrial ATP synthesis as measured by 31P-magnetic resonance spectroscopy (31P-MRS) from baseline up to 1 hour following study interventions

CONTACTS AND LOCATIONS:
Overall Officials: Russell Richardson, Ph.D., Principal Investigator — George E Wahlen VA Medical Center
Locations (1):
- George E Wahlen VA Medical Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No